CLINICAL TRIAL: NCT02093351
Title: An Open-Label, Non-randomised, Parallel Group, Multicentre, Phase I Study to Assess the Safety and Effect of Olaparib at Steady State on the Pharmacokinetics of the Anti-hormonal Agents Anastrozole, Letrozole and Tamoxifen at Steady State, and the Effect of the Anti-hormonal Agents on Olaparib, Following Administration in Patients With Advanced Solid Cancer
Brief Title: To Assess Safety and Effect of Olaparib on the Pharmacokinetics of Anastrozole, Letrozole & Tamoxifen, and Their Effect on Olaparib, in Patients With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D081CC00001
Record Dates: First submitted 2014-03-06; First posted 2014-03-21 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumours
Keywords: oncology, cancer, tumour, neoplasm, anticancer drug, pharmacokinetics, olaparib, anastrozole, tamoxifen, letrozole,
MeSH Terms: conditions — Neoplasms | interventions — olaparib; Tamoxifen; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 - Tamoxifen (Experimental): Olaparib-alone Steady state PK, Tamoxifen-alone steady state PK, Combined olaparib and Tamoxifen steady state PK.
  Interventions: Drug: Olaparib; Drug: Tamoxifen; Procedure: Pharmacokinetic sampling
- Cohort 2 - Anastrozole (Experimental): Olaparib-alone Steady state PK, Anastrozole-alone steady state PK, Combined olaparib and Anastrozole steady state PK.
  Interventions: Drug: Olaparib; Drug: Anastrozole; Procedure: Pharmacokinetic sampling
- Cohort 3 - Letrozole (Experimental): Olaparib-alone Steady state PK, Letrozole-alone steady state PK, Combined olaparib and Letrozole steady state PK.
  Interventions: Drug: Olaparib; Drug: Letrozole; Procedure: Pharmacokinetic sampling

INTERVENTIONS:
Drug: Olaparib — 2 x 150mg tablets, twice daily Day 1-5, and Day 27 onwards (Cohort 1), Day 20 onwards (Cohort 2) or Day 39 onwards (Cohort 3)
Drug: Tamoxifen — 60mg Tamoxifen once daily, Day 10 - Day 13; 20mg Tamoxifen once daily, Day 14 - Day 31
  Arms: Cohort 1 - Tamoxifen
Drug: Anastrozole — 1mg Anastrozole once daily Day 10 - Day 24
  Arms: Cohort 2 - Anastrozole
Drug: Letrozole — 2.5mg Letrozole once daily Day 10 - Day 43
  Arms: Cohort 3 - Letrozole
Procedure: Pharmacokinetic sampling — Blood sampling over 12-24 hour period for pharmacokinetic analysis

SUMMARY:
This is an open-label 2-part Phase I study in patients with advanced solid tumours. Part A of the study (mandatory) will assess the effect of olaparib on the pharmacokinetics (PK) of anastrozole, letrozole and tamoxifen and vice versa; Part B will allow patients (if eligible) continued access to olaparib after the PK phase and will provide additional safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures
2. Male or female aged ≥18 years
3. Histological or cytological confirmation of any malignant solid tumour in an advanced or metastatic setting who meet one of the criteria below:

   * Patients should be resistant or refractory to standard treatment if such treatment exists OR
   * Patients for which no suitable effective standard therapy exists OR
   * Patients with advanced breast cancer for whom anastrozole, letrozole or tamoxifen are indicated may also enter the study (postmenopausal breast cancer patients will be eligible for any of the cohorts; however, premenopausal breast cancer patients will be eligible for the tamoxifen cohort only).
4. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin (Hb) ≥10.0 g/dL with no blood transfusions in the past 28 days
   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) (except in the case of Gilbert's disease)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 x institutional ULN unless liver metastases are present, in which case they must be ≤5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
6. Patients must have a life expectancy ≥16 weeks
7. Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of Part A.

   Postmenopausal is defined as:
   * Age ≥ 60 years
   * Age <60 years and amenorrheic for 1 year or more in the absence of chemotherapy and/or hormonal treatment
   * Luteinising hormone (LH), follicle stimulating hormone (FSH) and plasma oestradiol levels in the postmenopausal range for women under 60 years
   * Radiation-induced oophorectomy with last menses >1 year ago
   * Or surgical sterilisation (bilateral oophorectomy or hysterectomy)
8. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment, and scheduled visits and examinations
9. Patients must be on stable concomitant medication regimen (with the exception of electrolyte supplements), defined as no change in medication or dose within 2 weeks prior to start of study treatment.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, its agents, and/or staff at the study site)
2. Previous enrolment in the present study
3. Exposure to an investigational product (IP) (including PARP inhibitor) within 30 days or 5 half lives (whichever is the longer) prior to enrolment
4. Prior chemotherapy within 3 weeks of study entry
5. Prior radiotherapy within 2 weeks of study entry
6. If prior endocrine treatment is given, adequate washout period is required: at least 2 weeks for anastrozole, at least 4 weeks for letrozole and at least 10 weeks for tamoxifen
7. Resting ECG with QTc >470 msec detected on 2 or more time points within a 24 hour period, or family history of long QT syndrome. If ECG demonstrates QTc >470 msec, patient will be eligible only if repeat ECG demonstrates QTc <470 msec.
8. Patients who are receiving inhibitors or inducers of CYP3A4 unless washed out prior to start of study treatment.
9. Persistent toxicities (Common Toxicity Criteria for Adverse Events [CTCAE] grade ≥2) caused by previous cancer therapy, excluding alopecia and/or CTCAE grade 2 peripheral neuropathy
10. Patients with myelodysplastic syndrome/acute myeloid leukaemia
11. Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery
12. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled seizures or active uncontrolled infection.
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with absorption of the study medication
14. Patients who have gastric, gastro-oesophageal, or oesophageal cancer
15. Pregnant or breastfeeding women
16. Patients with known active Hepatitis B or C, or human immunodeficiency virus (HIV).
17. Patients with a known hypersensitivity to olaparib (all cohorts), tamoxifen (Cohort 1) anastrozole (Cohort 2), letrozole (Cohort 3), or any of the excipients of these products.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsveta Milenkova, Study Director — AstraZeneca; Ruth Plummer, Principal Investigator — Sir Bobby Robson Cancer Trials Research Centre
Locations (14):
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Wilrijk
- Research Site, Herlev, Denmark
- Research Site, Bordeaux, France
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Utrecht
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

REFERENCES:
- [Derived] Plummer R, Verheul HM, De Vos FYFL, Leunen K, Molife LR, Rolfo C, Grundtvig-Sorensen P, De Greve J, Rottey S, Jerusalem G, Italiano A, Spicer J, Dirix L, Goessl C, Birkett J, Spencer S, Learoyd M, Bailey C, Dean E. Pharmacokinetic Effects and Safety of Olaparib Administered with Endocrine Therapy: A Phase I Study in Patients with Advanced Solid Tumours. Adv Ther. 2018 Nov;35(11):1945-1964. doi: 10.1007/s12325-018-0804-z. Epub 2018 Oct 15. PMID 30324586
- See also: Clinical Study Protocol REDACTED — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2882&filename=D081CC00001%20Clinical%20Study%20Protocol_REDACTED%20SECURED.PDF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 01 Sep 2014; last completed Part A: 28 Apr 2015. Last patient completed Part B: 27 Apr 2016. Part A assessed olaparib's effect on the pharmacokinetic (PK) parameters of anastrozole, letrozole and tamoxifen and vice versa; in Part B eligible patients received olaparib providing further safety data. Target accrual was met.
Pre-assignment Details: 79 patients were assigned to study treatment and received at least 1 dose of olaparib in Part A; 18 patients did not fulfil eligibility criteria. Part A of the study consisted of 3 treatment periods preceded by a screening period. There was a 4-day washout between the first two treatment periods.
Groups:
- Cohort 1 - Tamoxifen: In Part A, patients in Cohort 1 received olaparib 300 mg twice daily (bd) for 5 days in Treatment Period 1; tamoxifen 60 mg once daily (od) (loading dose) for 4 days then 20 mg od for 13 days (maintenance dose) in Treatment Period 2; and tamoxifen 20 mg od concomitantly with olaparib 300 mg bd for 5 days in Treatment Period 3.
- Cohort 2 - Anastrozole: In Part A, patients in Cohort 2 received olaparib 300 mg bd for 5 days in Treatment Period 1; anastrozole 1 mg od for 10 days in Treatment Period 2; and anastrozole 1 mg od concomitantly with olaparib 300 mg bd for 5 days in Treatment Period 3.
- Cohort 3 - Letrozole: In Part A, patients in Cohort 3 received olaparib 300 mg bd for 5 days in Treatment Period 1; letrozole 2.5 mg od for 29 days in Treatment Period 2; and letrozole 2.5 mg od concomitantly with olaparib 300 mg bd for 5 days in Treatment Period 3.
- Olaparib (Part B): In Part B, patients continued to receive olaparib 300 mg bd either as monotherapy or in combination with routine clinical regimes of letrozole, anastrazole or tamoxifen if deemed necessary by the investigator.
Period: Part A
Arm/Group | Cohort 1 - Tamoxifen | Cohort 2 - Anastrozole | Cohort 3 - Letrozole | Olaparib (Part B)
Started | 30 | 23 | 26 | 0
Completing Treatment Period 1 | 29 | 22 | 23 | 0
Completing Treatment Period 2 | 29 | 21 | 23 | 0
Completing Treatment Period 3 | 28 | 21 | 23 | 0
Completed | 28 | 21 | 23 | 0
Not Completed | 2 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Condition under investigation worsened | 2 | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Part B
Arm/Group | Cohort 1 - Tamoxifen | Cohort 2 - Anastrozole | Cohort 3 - Letrozole | Olaparib (Part B)
Started | 0 (Only the Olaparib (Part B) arm is applicable for this period.) | 0 (Only the Olaparib (Part B) arm is applicable for this period.) | 0 (Only the Olaparib (Part B) arm is applicable for this period.) | 69 (Eligible patients completing Part A entered Part B for continued access to olaparib.)
Completed | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 63
Not completed — Patient decision | 0 | 0 | 0 | 3
Not completed — Disease progression | 0 | 0 | 0 | 4
Not completed — Complete response | 0 | 0 | 0 | 1
Not completed — Adverse event + disease progression | 0 | 0 | 0 | 1
Not completed — Lack of therapeutic response | 0 | 0 | 0 | 12
Not completed — Condition under investigation worsened | 0 | 0 | 0 | 39
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled in Part A of the study and who received at least 1 dose of olaparib were included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Tamoxifen | Cohort 2 - Anastrozole | Cohort 3 - Letrozole | Total
Number analyzed (Participants) | 30 | 23 | 26 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (11.32) | 59.4 (11.68) | 64.0 (7.79) | 58.3 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 20 | 64
  Male | 4 | 5 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 20 | 64
  Male | 4 | 5 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 23 | 26 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 27 | 22 | 24 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Effect of Olaparib on Exposure to Tamoxifen - Cmax ss
Description: Tamoxifen, N-desmethyl tamoxifen (N-DMT) and endoxifen Cmax ss in the presence and absence of co-administered olaparib, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 5, 6, 8, 12 and 24 hours post-dose on Day 26 and Day 31
Population: The PK Analysis set included all patients who received a study drug dose and provided evaluable PK profiles for at least 1 treatment period in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Cohort 1 - Tamoxifen Alone (Treatment Period 2): Patients in Cohort 1 received tamoxifen 60 mg od from Day 10 to Day 13 (loading dose). From Day 14 to Day 26 patients received tamoxifen 20 mg od (maintenance dose). Blood sampling for PK analysis was taken on Day 26.
- Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3): Patients in Cohort 1 received tamoxifen 20 mg od concomitantly with olaparib 300 mg bd for 5 days from Day 27 to Day 31. Blood sampling for PK analysis was taken on Day 31.
Arm/Group | Cohort 1 - Tamoxifen Alone (Treatment Period 2) | Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3)
Number analyzed (Participants) | 24 | 18
mcg/mL
  PK analysis of tamoxifen | 130.3 (27.3) | 154.2 (34.9)
  PK analysis of N-DMT | 162.9 (28.0) | 149.1 (44.8)
  PK analysis of endoxifen | 5.923 (65.7) | 5.727 (61.2)
Statistical Analysis 1: Comparison: Cohort 1 - Tamoxifen Alone (Treatment Period 2) vs Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3); Analysis of tamoxifen PK parameters; Test type: Equivalence — If the 90% confidence interval (CI) for the tamoxifen treatment ratio falls within 0.7 to 1.43, olaparib can be considered to have had an effect on tamoxifen exposure that is unlikely to be clinically relevant; GLS Mean Ratio = 1.13, 90% CI 2-sided [1.06 to 1.22] — olaparib + tamoxifen vs. tamoxifen

2. Primary Outcome: Effect of Tamoxifen on Exposure to Olaparib - Cmax ss
Description: Olaparib Cmax ss in the presence and absence of co-administered tamoxifen, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Cohort 1 - Olaparib (Treatment Period 1): Patients received olaparib 300 mg bd from Day 1 to Day 4, and on Day 5 received olaparib 300 mg once (morning dose only). Blood sampling for PK analysis was taken on Day 5.
Arm/Group | Cohort 1 - Olaparib (Treatment Period 1) | Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3)
Number analyzed (Participants) | 27 | 19
mcg/mL | 9.456 (41.5) | 7.216 (43.6)
Statistical Analysis 1: Comparison: Cohort 1 - Olaparib (Treatment Period 1) vs Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — If the 90% CI for the olaparib treatment ratio falls within 0.7 to 1.43, tamoxifen can be considered to have had an effect on olaparib exposure that is unlikely to be clinically relevant; GLS Mean Ratio = 0.80, 90% CI 2-sided [0.71 to 0.90] — olaparib + tamoxifen vs. olaparib

3. Primary Outcome: Effect of Olaparib on Exposure to Anastrozole - Cmax ss
Description: Anastrozole maximum plasma concentration at steady state (Cmax ss) in the presence and absence of co-administered olaparib, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 19 and Day 24
Population: PK Analysis set included all patients who received a study drug dose and provided evaluable PK profiles for at least 1 treatment period in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (mcg/mL)
Groups:
- Cohort 2 - Anastrozole Alone (Treatment Period 2): Patients in Cohort 2 received anastrozole 1 mg od from Day 10 to Day 19. Blood sampling for PK analysis was taken on Day 19.
- Cohort 2 - Olaparib + Anastrozole (Treatment Period 3): Patients in Cohort 2 received anastrozole 1 mg od concomitantly with olaparib 300 mg bd for 5 days from Day 20 to Day 24. Blood sampling for PK analysis was taken on Day 24.
Arm/Group | Cohort 2 - Anastrozole Alone (Treatment Period 2) | Cohort 2 - Olaparib + Anastrozole (Treatment Period 3)
Number analyzed (Participants) | 20 | 19
micrograms per millilitre (mcg/mL) | 40.98 (36.2) | 35.83 (31.9)
Statistical Analysis 1: Comparison: Cohort 2 - Anastrozole Alone (Treatment Period 2) vs Cohort 2 - Olaparib + Anastrozole (Treatment Period 3); Analysis of anastrozole PK parameters; Test type: Equivalence — If the 90% CI for the anastrozole treatment ratio falls within 0.8 to 1.25, olaparib can be considered to have had little or no effect on anastrozole exposure; Geometric Least Squares (GLS) Mean Ratio = 0.90, 90% CI 2-sided [0.84 to 0.97] — olaparib + anastrozole vs. anastrozole

4. Primary Outcome: Effect of Anastrozole on Exposure to Olaparib - Cmax ss
Description: Olaparib Cmax ss in the presence and absence of co-administered anastrozole, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 24
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Cohort 2 - Olaparib (Treatment Period 1): Patients received olaparib 300 mg bd from Day 1 to Day 4, and on Day 5 received olaparib 300 mg once (morning dose only). Blood sampling for PK analysis was taken on Day 5.
Arm/Group | Cohort 2 - Olaparib (Treatment Period 1) | Cohort 2 - Olaparib + Anastrozole (Treatment Period 3)
Number analyzed (Participants) | 22 | 20
mcg/mL | 9.490 (34.3) | 8.256 (39.9)
Statistical Analysis 1: Comparison: Cohort 2 - Olaparib (Treatment Period 1) vs Cohort 2 - Olaparib + Anastrozole (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — If the 90% CI for the olaparib treatment ratio falls within 0.7 to 1.43, anastrozole can be considered to have had an effect on olaparib exposure that is unlikely to be clinically relevant; GLS Mean Ratio = 0.94, 90% CI 2-sided [0.84 to 1.04] — olaparib + anastrozole vs. olaparib

5. Primary Outcome: Effect of Olaparib on Exposure to Letrozole - Cmax ss
Description: Letrozole Cmax ss in the presence and absence of co-administered olaparib, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 38 and Day 43
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Cohort 3 - Letrozole Alone (Treatment Period 2): Patients in Cohort 3 received letrozole 2.5 mg od from Day 10 to Day 38. Blood sampling for PK analysis was taken on Day 38.
- Cohort 3 - Olaparib + Letrozole (Treatment Period 3): Patients in Cohort 3 received letrozole 2.5 mg od concomitantly with olaparib 300 mg bd for 5 days from Day 39 to Day 43. Blood sampling for PK analysis was taken on Day 43.
Arm/Group | Cohort 3 - Letrozole Alone (Treatment Period 2) | Cohort 3 - Olaparib + Letrozole (Treatment Period 3)
Number analyzed (Participants) | 23 | 23
mcg/mL | 118.9 (32.6) | 111.8 (30.4)
Statistical Analysis 1: Comparison: Cohort 3 - Letrozole Alone (Treatment Period 2) vs Cohort 3 - Olaparib + Letrozole (Treatment Period 3); Analysis of letrozole PK parameters; Test type: Equivalence — If the 90% CI for the letrozole treatment ratio falls within 0.8 to 1.25, olaparib can be considered to have had little or no effect on letrozole exposure; GLS Mean Ratio = 0.94, 90% CI 2-sided [0.91 to 0.98] — olaparib + letrozole vs. letrozole

6. Primary Outcome: Effect of Letrozole on Exposure to Olaparib - Cmax ss
Description: Olaparib Cmax ss in the presence and absence of co-administered letrozole, and associated Cmax ss treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 43
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Cohort 3 - Olaparib (Treatment Period 1): Patients received olaparib 300 mg bd from Day 1 to Day 4, and on Day 5 received olaparib 300 mg once (morning dose only). Blood sampling for PK analysis was taken on Day 5.
Arm/Group | Cohort 3 - Olaparib (Treatment Period 1) | Cohort 3 - Olaparib + Letrozole (Treatment Period 3)
Number analyzed (Participants) | 22 | 23
mcg/mL | 10.05 (30.2) | 10.48 (33.6)
Statistical Analysis 1: Comparison: Cohort 3 - Olaparib (Treatment Period 1) vs Cohort 3 - Olaparib + Letrozole (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — If the 90% CI for the olaparib treatment ratio falls within 0.7 to 1.43, letrozole can be considered to have had an effect on olaparib exposure that is unlikely to be clinically relevant; GLS Mean Ratio = 1.09, 90% CI 2-sided [0.99 to 1.21] — olaparib + letrozole vs. olaparib

7. Primary Outcome: Effect of Olaparib on Exposure to Tamoxifen - AUC0-τ
Description: Tamoxifen, N-DMT and endoxifen AUC0-τ, in the presence and absence of co-administered olaparib, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 5, 6, 8, 12 and 24 hours post-dose on Day 26 and Day 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram x hour/millilitre (mcg*h/mL)
Arm/Group | Cohort 1 - Tamoxifen Alone (Treatment Period 2) | Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3)
Number analyzed (Participants) | 24 | 18
microgram x hour/millilitre (mcg*h/mL)
  PK analysis of tamoxifen | 2233 (31.9) | 2751 (28.9)
  PK analysis of N-DMT | 3189 (28.8) | 2955 (37.3)
  PK analysis of endoxifen | 119.3 (66.1) | 115.8 (64.8)
Statistical Analysis 1: Comparison: Cohort 1 - Tamoxifen Alone (Treatment Period 2) vs Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3); Analysis of tamoxifen PK parameters; Test type: Equivalence — If the 90% CI for the tamoxifen treatment ratio falls within 0.7 to 1.43, olaparib can be considered to have had an effect on tamoxifen exposure that is unlikely to be clinically relevant; GLS Mean Ratio = 1.16, 90% CI 2-sided [1.11 to 1.21] — olaparib + tamoxifen vs. tamoxifen

8. Primary Outcome: Effect of Tamoxifen on Exposure to Olaparib - AUC0-τ
Description: Olaparib AUC0-τ, in the presence and absence of co-administered tamoxifen, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 31
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Cohort 1 - Olaparib (Treatment Period 1) | Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3)
Number analyzed (Participants) | 26 | 18
mcg*h/mL | 62.12 (51.6) | 42.27 (60.6)
Statistical Analysis 1: Comparison: Cohort 1 - Olaparib (Treatment Period 1) vs Cohort 1 - Olaparib + Tamoxifen (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; GLS Mean Ratio = 0.73, 90% CI 2-sided [0.63 to 0.84] — olaparib + tamoxifen vs. olaparib

9. Primary Outcome: Effect of Olaparib on Exposure to Anastrozole - AUC0-τ
Description: Anastrozole Area under plasma concentration-time curve over the dosing interval at steady state (AUC0-τ), in the presence and absence of co-administered olaparib, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 19 and Day 24
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Cohort 2 - Anastrozole Alone (Treatment Period 2) | Cohort 2 - Olaparib + Anastrozole (Treatment Period 3)
Number analyzed (Participants) | 20 | 19
mcg*h/mL | 696.8 (36.6) | 582.5 (31.6)
Statistical Analysis 1: Comparison: Cohort 2 - Anastrozole Alone (Treatment Period 2) vs Cohort 2 - Olaparib + Anastrozole (Treatment Period 3); Analysis of anastrozole PK parameters; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GLS Mean Ratio = 0.86, 90% CI 2-sided [0.80 to 0.93] — olaparib + anastrozole vs. anastrozole

10. Primary Outcome: Effect of Anastrozole on Exposure to Olaparib - AUC0-τ
Description: Olaparib AUC0-τ, in the presence and absence of co-administered anastrozole, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 24
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Cohort 2 - Olaparib (Treatment Period 1) | Cohort 2 - Olaparib + Anastrozole (Treatment Period 3)
Number analyzed (Participants) | 21 | 19
mcg*h/mL | 55.49 (53.8) | 44.33 (63.6)
Statistical Analysis 1: Comparison: Cohort 2 - Olaparib (Treatment Period 1) vs Cohort 2 - Olaparib + Anastrozole (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GLS Mean Ratio = 0.89, 90% CI 2-sided [0.76 to 1.05] — olaparib + anastrozole vs. olaparib

11. Primary Outcome: Effect of Olaparib on Exposure to Letrozole - AUC0-τ
Description: Letrozole AUC0-τ, in the presence and absence of co-administered olaparib, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 38 and Day 43
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Cohort 3 - Letrozole Alone (Treatment Period 2) | Cohort 3 - Olaparib + Letrozole (Treatment Period 3)
Number analyzed (Participants) | 23 | 23
mcg*h/mL | 2292 (36.7) | 2167 (38.0)
Statistical Analysis 1: Comparison: Cohort 3 - Letrozole Alone (Treatment Period 2) vs Cohort 3 - Olaparib + Letrozole (Treatment Period 3); Analysis of letrozole PK parameters; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; GLS Mean Ratio = 0.95, 90% CI 2-sided [0.91 to 0.99] — olaparib + letrozole vs. letrozole

12. Primary Outcome: Effect of Letrozole on Exposure to Olaparib - AUC0-τ
Description: Olaparib AUC0-τ, in the presence and absence of co-administered letrozole, and associated AUC0-τ treatment ratios
Time Frame: Pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on Day 5 and Day 43
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Cohort 3 - Olaparib (Treatment Period 1) | Cohort 3 - Olaparib + Letrozole (Treatment Period 3)
Number analyzed (Participants) | 22 | 23
mcg*h/mL | 61.77 (43.2) | 67.82 (44.1)
Statistical Analysis 1: Comparison: Cohort 3 - Olaparib (Treatment Period 1) vs Cohort 3 - Olaparib + Letrozole (Treatment Period 3); Analysis of olaparib PK parameters; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; GLS Mean Ratio = 1.15, 90% CI 2-sided [1.07 to 1.25] — olaparib + letrozole vs. olaparib

ADVERSE EVENTS:
Time Frame: For Part A, adverse events (AEs) were collected from the date of first dose up to last dose of study medication in Part A for patients continuing to Part B, or up to 30 days after last dose for patients who did not enter Part B (up to approximately 2 months). For Part B, AEs were collected from date of first dose in Part B up to 30 days after last dose (up to approximately 18 months).
Description: AE data is reported as treatment-emergent AEs. Each Part A cohort received treatment over 3 Treatment Periods. There was a washout period of 4 days between Treatment Periods 1 and 2, and no washout period between Treatment Periods 2 and 3. MedDRA v18.1 was used for Part B.
Arm/Group | Cohort 1 - Tamoxifen | Cohort 2 - Anastrozole | Cohort 3 - Letrozole | Olaparib (Part B)
All-Cause Mortality (participants affected / at risk) | 1/30 | 1/23 | 1/26 | 1/69
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/23 | 0/26 | 22/69
Other Adverse Events (participants affected / at risk) | 27/30 | 20/23 | 20/26 | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Tamoxifen (N=30) | Cohort 2 - Anastrozole (N=23) | Cohort 3 - Letrozole (N=26) | Olaparib (Part B) (N=69)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8)
Klebsiella Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior Vena Cava Occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Tamoxifen (N=30) | Cohort 2 - Anastrozole (N=23) | Cohort 3 - Letrozole (N=26) | Olaparib (Part B) (N=69)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 3 (3) | 3 (3) | 18 (27)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (7)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 10 (13)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (4) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (5) | 12 (13)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 16 (22) | 7 (12) | 11 (13) | 28 (32)
Vomiting (Gastrointestinal disorders) | 6 (9) | 4 (4) | 4 (5) | 22 (34)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (6)
Fatigue (General disorders) | 12 (13) | 6 (7) | 9 (10) | 30 (36)
Non-Cardiac Chest Pain (General disorders) | 2 (3) | 0 (0) | 3 (3) | 5 (6)
Oedema Peripheral (General disorders) | 2 (2) | 2 (3) | 2 (2) | 7 (8)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 3 (3)
Blood Creatinine Increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 3 (4) | 13 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4) | 1 (1) | 8 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 6 (6)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (5) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 9 (12)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 9 (9)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 4 (4) | 12 (21)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4) | 1 (1) | 18 (21)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 2 (2) | 3 (4)
Hot Flush (Vascular disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Vaginal Discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (6)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 1 (1) | 10 (10)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 9 (9)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Gamma-glutamyltransferase Increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6)

LIMITATIONS AND CAVEATS:
At the end of Part B, the continued access phase (CAP) allowed patients to continue to receive olaparib if deriving clinical benefit. No clinical data was databased during the CAP, thus AE data is presented to the end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No